CLINICAL TRIAL: NCT07351422
Title: Investigating Management, Perspectives and Attitudes Towards Care in Takayasu Arteritis
Acronym: TAK-IMPACT
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 25-EMREC-064
Record Dates: First submitted 2025-11-14; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Takayasu Arteritis; Takayasu Arteritis (TAK)
MeSH Terms: conditions — Takayasu Arteritis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Takayasu Arteritis
  Interventions: Other: Questionnaire
- Physicians Involved in the Management of Patients with Takayasu Arteritis
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — An online annoymous questionnaire consisting of short-answer and multiple-choice questions

SUMMARY:
This study aims to understand the experiences of patients with Takayasu arteritis (TAK) and how physicians manage the condition. To achieve this, two separate questionnaires will be conducted: one for patients and one for physicians.

DETAILED DESCRIPTION:
This study aims to investigate the experiences and perceptions of patients with Takayasu arteritis regarding their disease, as well as the perspectives of physicians regarding the management and treatment of these patients.

Patients with TAK will be invited to complete an anonymous online (Online Surveys) questionnaire, which will take approximately 25 minutes and will consist of multiple-choice and short-answer questions. The questionnaire will ask about their experience with the condition, symptoms, treatments they have received, and any concerns or priorities they have regarding their care.

Physicians who treat TAK will also be invited to complete a separate online questionnaire, taking around 15 minutes and also consisting of multiple-choice and short-answer questions. This will explore how they diagnose and manage TAK, their choice of treatments, and any challenges they face in treating the condition

ELIGIBILITY:
Inclusion Criteria:

For the patient questionnaire:

* Age ≥ 18 years
* A formal diagnosis of TAK

For the physician questionnaire

• A physician involved in the management/decision-making for patients diagnosed with TAK

Exclusion Criteria:

For the patient questionnaire:

* Age < 18 years
* Lack of a formal diagnosis of TAK
* Patients without mental capacity or willingness to provide informed consent
* Not UK based

For the physician questionnaire

* Not involved in the management/ decision making for patients diagnosed with TAK
* Not willing to take part
* Not UK based

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are UK-based
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Patient Perspective | Day 1
  To understand the lived experiences of individuals with TAK, including their symptoms, health status post-diagnosis, treatment priorities, and concerns.
  The questionnaire covers the following topics:
  * Basic background information
  * Living with Takayasu arteritis
  * Changes to health since diagnosis
  * Physical activity and exercise habits- measured by the International Physical Activity Questionnaire (IPAQ)
  * Smoking history
  * Mental well-being- measured by the EQ-5D instrument
  * Nutrition and diet
  * Personal views and priorities on management
Physician Perspective | Day 1
  To evaluate current clinical management strategies for TAK, identify treatment priorities, and highlight areas of unmet need in clinical practice.
  The physician questionnaire covers the following topics:
  * Clinical background and experience with TAK patients
  * Diagnostic and treatment strategies for TAK
  * Consideration of cardiovascular disease risk in TAK management
  * Physician priorities and unmet needs of management

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No